CLINICAL TRIAL: NCT01541982
Title: Virtual Autopsy for Quality Control on Intensive Care Medicine
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: VA-2 Quality Control
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Value of Virtual Autopsy for Quality Control in Icu

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- virtual and classic autopsy: "Goldstandard": A group of patients in which virtual and classic autopsy is performed.
- virtual autopsy only: "Intervention": A group of patients in which for various reasons virtual autopsy only is performed.

SUMMARY:
The study aimed to compare CT-based virtual autopsy with classic autopsy as a tool for quality control in intensive care medicine.

DETAILED DESCRIPTION:
The study aimed to compare CT-based virtual autopsy with classic autopsy as a tool for quality control in intensive care medicine. Especially with respect to complications during intervention like catheter pacement.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* all patients dying in the icu during the study period

Exclusion Criteria:

* relatives refuse participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients dying in the icu
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Wichmann, MD, Principal Investigator — Department of Intensive Care Medicine, University Medical Center Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - Department of Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg

REFERENCES:
- [Derived] Wichmann D, Heinemann A, Zahler S, Vogel H, Hopker W, Puschel K, Kluge S. Prospective study of device-related complications in intensive care unit detected by virtual autopsy. Br J Anaesth. 2018 Jun;120(6):1229-1236. doi: 10.1016/j.bja.2018.02.031. Epub 2018 Apr 4. PMID 29793590